CLINICAL TRIAL: NCT05141890
Title: Probiotics for Inflammation in Pediatric Chronic Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Keri Hainsworth, Associate Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1679041
Record Dates: First submitted 2021-11-17; First posted 2021-12-02 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain; Body Mass Index >=85th Percentile
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotic (Experimental): Participants will be given the probiotic supplement Lp299v. The supplement is taken by mouth in the form of capsules. Participants will undergo a screening visit. After 7-11 weeks of taking Lp299v, they will return for their final visit. Blood will be drawn before and after the 7- 11 week intervention.
  Interventions: Dietary Supplement: Lactobacillus Plantarum

INTERVENTIONS:
Dietary Supplement: Lactobacillus Plantarum — Dietary Supplement: Lp299v. Lp299v is a commercially available probiotic supplement manufactured and distributed by Next Foods.
  Other Names: Lp299v

SUMMARY:
To examine benefits of a probiotic for youth with chronic pain and a Body Mass Index >=85th percentile.

DETAILED DESCRIPTION:
The purpose of the current study: (1) examine whether a 7-11 week supplement of a single-strain probiotic (Lactobascillus Plantarum, Lp299v) reduces systemic inflammation; (2) determine whether reductions in systemic inflammation will correlate with reductions in pain, disability, mood impairment and changes in mechanical pain threshold and mechanical pain sensitization; (3) Explore whether reductions in systemic inflammation will correlate with reductions in other outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female biological sex
2. 13-17 years of age
3. Body Mass Index ≥85th percentile for sex and age

Exclusion Criteria:

1. Probiotic (or prebiotic) supplement use or antibiotic use within the past month
2. Chronic inflammatory or autoimmune disease with the exception of well-controlled hypothyroidism or intermittent or mild persistent asthma not requiring the use of daily inhaled steroids
3. Patients who have had a poor response to blood draw or immunizations in the past
4. Chronic use of medications known to alter gastrointestinal function or inflammation (e.g. metformin, non-steroidal anti-inflammatory medications)
5. Any condition that, in the investigator's opinion, may compromise study participation or may confound the interpretation of the study results
6. Use of illicit drugs
7. Females who are pregnant or lactating

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in systemic inflammation - CRP | 7-11 weeks
  Change in circulating C-Reactive Protein after 8 weeks of probiotic supplement.

SECONDARY OUTCOMES:
Change in Worst Pain intensity | 7-11 weeks
  Change in worst pain intensity (based on a 0-10 numeric rating scale) over the past 2 weeks after 7-11 weeks of probiotic supplement.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No